CLINICAL TRIAL: NCT04321122
Title: Observation on the Clinical Safety and Efficacy of UCP (Ultrasound Cyclo Plasty) in the Treatment of Chinese Patients With Primary Open-angle Glaucoma
Brief Title: UCP (Ultrasound Cyclo Plasty) in the Treatment of Chinese Patients With Primary Open-angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018QXPJ005
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-06

CONDITIONS: Glaucoma; Glaucoma, Primary Open Angle
Keywords: Primary open-angle glaucoma; UCP(ultrasound cyclo plasty); Efficacy and Safety
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound cyclo plasty(UCP) (Experimental): Ultrasound cyclo plasty treatment for primary open-angle glaucoma patients.
  Interventions: Procedure: ultrasound cyclo plasty

INTERVENTIONS:
Procedure: ultrasound cyclo plasty — The "ultrasonic glaucoma treatment instrument" produced by French EYE TECH CARE company is referred to as EyeOP1.It uses high-intensity focused ultrasound technique to make target part of the ciliary coagulative necrosis, reduce the production of aqueous humor and thereby lower the intraocular pressure. EyeOP1 is ergonomic and suitable for the human eye, making the treatment process more accurate, simple and fast.
  Other Names: UCP

SUMMARY:
Traditional ciliary body photocoagulation treatment uses the photocoagulation of long-wavelength laser to destroy the ciliary body tissue that can produce aqueous humor. Therefore, it is a kind of palliative treatment which has proved efficacy but causes great pain to patients. The "ultrasonic glaucoma treatment instrument" produced by French EYE TECH CARE company is referred to as EyeOP1. It uses high-intensity focused ultrasound technique to make target part of the ciliary coagulative necrosis, reduce the production of aqueous humor and thereby lower the intraocular pressure. EyeOP1 is ergonomic and suitable for the human eye, making the treatment process more accurate, simple and fast.

DETAILED DESCRIPTION:
1. Efficacy: 1. Main objective: (1)Assess the decrease in postoperative intraocular pressure from baseline and evaluate the final results (the percentage of patients whose conditions have significant improved and the variation of the percentage of median intraocular pressure. (2)Assess the amount of medication after surgery.
2. Secondary goals:(1) Compare median intraocular pressure with baseline at each postoperative follow-up and access the variation of median intraocular pressure from baseline at each postoperative follow-up. (2) Count the number of intraocular pressure lowering drugs at each postoperative follow-up.

b.Safety: Investigate the incidence of all device-related(or procedure-related) adverse events during the study (intraoperative and postoperative follow-up).

ELIGIBILITY:
Inclusion Criteria:

* The target eye was diagnosed as primary open-angle glaucoma; diagnostic criteria: IOP(intraocular pressure)≥ 21, open angle, typical glaucoma visual field and optic disc damage;
* Patients treated with glaucoma medications cannot control intraocular pressure effectively;
* Patients with 21mmHg ≤ IOP ≤ 30mmHg;
* VA(visual acuity)≥HM(hand motions);
* Patients that have failed conventional glaucoma surgery (trabeculectomy) or are not suitable for surgery;
* Patients who have not received intraocular surgery or laser treatment 90 days before receiving HIFU;
* Aged from 18 to 90 years old;
* Sign informed consent and be willing to provide visit data;

Exclusion Criteria:

* Either eye have any infections two weeks before the surgery;
* The target eye has history of ciliary surgery, intraocular or retrobulbar tumor;
* The target eye is neovascular glaucoma;
* The target eye is aphakic eye;
* Anterior anatomical abnormalities cause scleral expansion or ciliary body ectopic;
* Non-glaucoma intraocular diseases that affect intraocular pressure;
* Within 30 days, the patient participated in or was simultaneously included in other clinical trials;
* Patients during pregnancy or lactation;
* Any systemic disease that may affect patient follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-12 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-06-12 (Estimated)

PRIMARY OUTCOMES:
IOP(intraocular pressure) | 6 months after surgery
  To evaluate the success rate of IOP control at 6 months after UCP(5mmHg≤IOP≤21mmHg, and at least 20% lower than the baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Ge, M.D,Ph.D, Study Chair — Zhognshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The archived documents and materials are not loaned. If the management department needs to access the original data, it should be agreed by the PI of the project.